CLINICAL TRIAL: NCT02452047
Title: A Phase III, Randomized, Double-Blind, Active Comparator-Controlled Clinical Trial to Estimate the Efficacy and Safety of Imipenem/Cilastatin/Relebactam (MK-7655A) Versus Colistimethate Sodium + Imipenem/Cilastatin in Subjects With Imipenem-Resistant Bacterial Infection
Brief Title: Efficacy and Safety of Imipenem+Cilastatin/Relebactam (MK-7655A) Versus Colistimethate Sodium+Imipenem+Cilastatin in Imipenem-Resistant Bacterial Infection (MK-7655A-013)
Acronym: RESTORE-IMI 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7655A-013; 2015-000066-62 (EudraCT Number); 163367 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — imipenem, cilastatin and relebactam; colistinmethanesulfonic acid; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Imipenem+Cilastatin/Relebactam (Experimental): Participants will be stratified by infection type (HABP/VABP, cIAI, and cUTI) and randomized to receive imipenem+cilastatin/relebactam intravenous (IV) infusion once every 6 hours and placebo for colistimethate sodium IV infusion once every 12 hours for 5 to 21 days for cIAI and cUTI or for 7 to 21 days for HABP or VABP. Treatment durations >21 days may be approved by the Sponsor for participants requiring longer treatment duration.
  Interventions: Drug: Imipenem+Cilastatin/Relebactam; Drug: Placebo to CMS
- Group 2: Colistimethate sodium + Imipenem+Cilastatin (Active Comparator): Participants will be stratified by infection type (HABP/VABP, cIAI, and cUTI) and randomized to receive colistimethate sodium IV infusion once every 12 hours and imipenem+cilastatin IV infusion once every 6 hours for 5 to 21 days for cIAI and cUTI or for 7 to 21 days for HABP or VABP. Treatment durations >21 days may be approved by the Sponsor for participants requiring longer treatment duration.
  Interventions: Drug: Colistimethate sodium (CMS); Drug: Imipenem+Cilastatin
- Group 3: Imipenem+Cilastatin/Relebactam (Experimental): Participants with documented imipenem-resistant and colistin-resistant bacterial infections may be eligible to receive open-label imipenem+cilastatin/relebactam IV infusion once every 6 hours for 5 to 21 days for cIAI and cUTI or for 7 to 21 days for HABP or VABP. Treatment durations >21 days may be approved by the Sponsor for participants requiring longer treatment duration.
  Interventions: Drug: Imipenem+Cilastatin/Relebactam

INTERVENTIONS:
Drug: Imipenem+Cilastatin/Relebactam — Imipenem+Cilastatin/Relebactam 200/100 mg to 500/250 mg, depending on renal function, IV infusion once every 6 hours
  Other Names: MK-7655A
  Arms: Group 1: Imipenem+Cilastatin/Relebactam; Group 3: Imipenem+Cilastatin/Relebactam
Drug: Colistimethate sodium (CMS) — Colistimethate base activity 300 mg (~720 mg CMS) IV infusion loading dose, followed by colistimethate base activity 75 mg to 150 mg (~180 to 360 mg CMS), depending on renal function, once every 12 hours
  Arms: Group 2: Colistimethate sodium + Imipenem+Cilastatin
Drug: Imipenem+Cilastatin — Imipenem+cilastatin 200 mg to 500 mg, depending on renal function, IV infusion once every 6 hours
  Arms: Group 2: Colistimethate sodium + Imipenem+Cilastatin
Drug: Placebo to CMS — Placebo to CMS IV infusion once every 12 hours
  Arms: Group 1: Imipenem+Cilastatin/Relebactam

SUMMARY:
The study will evaluate the efficacy and safety of imipenem+cilastatin/relebactam (MK-7655A) versus colistimethate sodium+imipenem+cilastatin in the treatment of imipenem-resistant bacterial infections. Infections evaluated in the study will be hospital-acquired bacterial pneumonia (HABP), ventilator-associated bacterial pneumonia (VABP), complicated intra-abdominal infection (cIAI), and complicated urinary tract infection (cUTI).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization that requires treatment with IV antibiotic therapy for a new, persistent or progressing bacterial infection involving at least 1 of 3 primary infection types (HABP, VABP, cIAI, or cUTI)
* Positive culture data from the primary infection-site specimen collected within 1 week of study entry. At least one of the suspected causative pathogens from the specimen meets all of the following: 1) identified as a Gram-negative bacterium, 2) culture-confirmed imipenem resistance (and colistin resistance for Group 3 only), 3) culture-confirmed susceptibility to imipenem/relebactam and to colistin (for Groups 1 and 2 only)
* Not of reproductive potential, or of reproductive potential and agrees to avoid becoming pregnant or impregnating a partner by complying with one of the following: 1) practice abstinence, or 2) use of acceptable contraception during heterosexual activity

Exclusion Criteria:

* Concurrent infection (endocarditis, osteomyelitis, meningitis, prosthetic joint infection, disseminated fungal infection, or active pulmonary tuberculosis) that would interfere with evaluation of the response to the study antibiotics
* Received treatment with any form of systemic colistin for >24 hours within 72 hours before initiation of study drug (for Groups 1 and 2 only)
* HABP or VABP caused by an obstructive process
* cUTI which meets any of the following: 1) complete obstruction of any portion of the urinary tract, 2) known ileal loop, 3) intractable vesico-ureteral reflux, 4) presence of an indwelling urinary catheter which cannot be removed at study entry
* History of serious allergy, hypersensitivity, or any serious reaction to listed antibiotics (per-protocol)
* Female who is pregnant or is expecting to conceive (or a male partner of a female who is expecting to conceive), is breastfeeding, or plans to breastfeed before completion of the study
* Anticipated treatment with any of the following during the study: valproic acid or divalproex sodium, or concomitant systemic (e.g. IV, oral or inhaled) antimicrobial agents with known Gram-negative bacterial coverage
* Currently undergoing hemodialysis or peritoneal dialysis
* Participated or anticipates participating in any other clinical study involving administration of investigational medication up to 30 days before screening or during the course of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08-21 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Brown ML, Motsch J, Kaye KS, File TM, Boucher HW, Vendetti N, Aggrey A, Joeng HK, Tipping RW, Du J, DePestel DD, Butterton JR, Paschke A. Evaluation of Renal Safety Between Imipenem/Relebactam and Colistin Plus Imipenem in Patients With Imipenem-Nonsusceptible Bacterial Infections in the Randomized, Phase 3 RESTORE-IMI 1 Study. Open Forum Infect Dis. 2020 Feb 19;7(3):ofaa054. doi: 10.1093/ofid/ofaa054. eCollection 2020 Mar. PMID 32154325
- [Derived] Kaye KS, Boucher HW, Brown ML, Aggrey A, Khan I, Joeng HK, Tipping RW, Du J, Young K, Butterton JR, Paschke A. Comparison of Treatment Outcomes between Analysis Populations in the RESTORE-IMI 1 Phase 3 Trial of Imipenem-Cilastatin-Relebactam versus Colistin plus Imipenem-Cilastatin in Patients with Imipenem-Nonsusceptible Bacterial Infections. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e02203-19. doi: 10.1128/AAC.02203-19. Print 2020 Apr 21. PMID 32094127
- [Derived] Motsch J, Murta de Oliveira C, Stus V, Koksal I, Lyulko O, Boucher HW, Kaye KS, File TM, Brown ML, Khan I, Du J, Joeng HK, Tipping RW, Aggrey A, Young K, Kartsonis NA, Butterton JR, Paschke A. RESTORE-IMI 1: A Multicenter, Randomized, Double-blind Trial Comparing Efficacy and Safety of Imipenem/Relebactam vs Colistin Plus Imipenem in Patients With Imipenem-nonsusceptible Bacterial Infections. Clin Infect Dis. 2020 Apr 15;70(9):1799-1808. doi: 10.1093/cid/ciz530. PMID 31400759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with hospital-acquired bacterial pneumonia (HABP), ventilator-associated bacterial pneumonia (VABP), complicated intra-abdominal infection (cIAI), or complicated urinary tract infection (cUTI) were recruited at 35 study centers in 17 countries.
Groups:
- Group 1: Imipenem+Cilastatin/Relebactam: Participants with HABP, VABP, cIAI, or cUTI caused by imipenem-nonsusceptible but imipenem/relebactam- and colistin-susceptible pathogens were randomized to receive imipenem+cilastatin/relebactam IV infusion once every 6 hours and placebo for colistimethate sodium IV infusion once every 12 hours for 5 to 21 days (cIAI and cUTI) or for 7 to 21 days (HABP or VABP).
- Group 2: Colistimethate Sodium + Imipenem+Cilastatin: Participants with HABP, VABP, cIAI, or cUTI caused by imipenem-nonsusceptible but imipenem/relebactam- and colistin-susceptible pathogens were randomized to receive colistimethate sodium IV infusion once every 12 hours and imipenem+cilastatin IV infusion once every 6 hours for 5 to 21 days (cIAI and cUTI) or for 7 to 21 days (HABP or VABP).
- Group 3: Open-Label Imipenem+Cilastatin/Relebactam: Participants with HABP, VABP, cIAI, or cUTI caused by imipenem- and colistin-nonsusceptible pathogens received open-label imipenem+cilastatin/relebactam IV infusion once every 6 hours for 5 to 21 days (cIAI and cUTI) or for 7 to 21 days (HABP or VABP).
Period: Overall Study
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Started | 31 | 16 | 3
Completed | 27 | 11 | 1
Not Completed | 4 | 5 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Death | 1 | 3 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam | Total
Number analyzed (Participants) | 31 | 16 | 3 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (16.5) | 62.8 (14.9) | 50.0 (23.1) | 57.9 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 2 | 19
  Male | 20 | 10 | 1 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 26 | 15 | 3 | 44
  More than one race | 4 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Favorable Overall Response (FOR)
Description: The percentage of participants with FOR was determined for Groups 1 and 2. FOR was determined based on clinically relevant outcomes for the primary site of infection as follows: HABP/VABP: survival through Day 28; cIAI: favorable clinical response (all pretherapy symptoms of index infection resolved with no evidence of resurgence, no additional antibiotic therapy required, and no unplanned surgical or percutaneous drainage procedures) at Day 28; cUTI: favorable composite clinical response (all pretherapy symptoms of index infection resolved with no evidence of resurgence, no additional antibiotic therapy required) and microbiological response (urine culture shows sustained eradication of the baseline uropathogen [e.g., ≥10^5 CFU/mL at study entry is reduced to <10^4 CFU/mL]) at Early Follow-up (EFU).
Time Frame: Up to Day 30 (up to 9 days after completing study treatment)
Population: Participants in Groups 1 and 2 who received ≥1 dose of each trial drug within a given IV treatment regimen, and who had a baseline bacterial pathogen that met inclusion criteria, are included. As per protocol, efficacy data from open-label Group 3 was considered exploratory and not included in the comparative analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 21 | 10 | 0
Percentage of Participants | 71.4 [49.8 to 86.4] | 70.0 [39.2 to 89.7] |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in FOR % = -7.3, 90% CI 2-sided [-27.5 to 21.4] — Stratified Miettinen & Nurminen method by infection type

2. Primary Outcome: Percentage of Participants With ≥1 Adverse Events (AEs)
Description: The percentage of participants in Groups 1, 2, and 3 experiencing ≥1 AEs during treatment and 14-day follow-up was determined. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Statistical analysis included only Groups 1 and 2 as indicated by the protocol.
Time Frame: Up to Day 35 (up to 14 days after completing study treatment)
Population: All participants in Groups 1, 2, and 3 who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 31 | 16 | 3
Percentage of Participants | 71.0 | 81.3 | 100.0
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in AE % = -10.3, 95% CI 2-sided [-33.1 to 18.0] — Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants With ≥1 Serious Adverse Events (SAEs)
Description: The percentage of participants in Groups 1, 2, and 3 experiencing ≥1 SAEs during treatment and 14-day follow-up was determined. An SAE is any untoward medical occurrence that, at any dose, results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant injury/incapacity; is a congenital anomaly/birth defect; or is an other important medical event. Statistical analysis included only Groups 1 and 2 as indicated by the protocol.
Time Frame: Up to Day 35 (up to 14 days after completing study treatment)
Population: All participants in Groups 1, 2, and 3 who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 31 | 16 | 3
Percentage of Participants | 9.7 | 31.3 | 100.0
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in SAE % = -21.6, 95% CI 2-sided [-47.8 to 1.3] — Miettinen & Nurminen method

4. Primary Outcome: Percentage of Participants With ≥1 Drug-Related AEs
Description: The percentage of participants in Groups 1, 2, and 3 experiencing ≥1 drug-related AEs during treatment and 14-day follow-up was determined. A drug-related AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, and considered by the investigator to be related to the study intervention. Statistical analysis included only Groups 1 and 2 as indicated by the protocol.
Time Frame: Up to Day 35 (up to 14 days after completing study treatment)
Population: All participants in Groups 1, 2, and 3 who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 31 | 16 | 3
Percentage of Participants | 16.1 | 31.3 | 33.3
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in drug-related AE % = -15.1, 95% CI 2-sided [-42.3 to 9.2] — Miettinen & Nurminen method

5. Primary Outcome: Percentage of Participants With ≥1 Drug-Related SAEs
Description: The percentage of participants in Groups 1, 2, and 3 experiencing ≥1 drug-related SAEs during treatment and 14-day follow-up was determined. A drug-related SAE is any untoward medical occurrence that, at any dose, results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant injury/incapacity; is a congenital anomaly/birth defect; or is an other important medical event, that is considered by the investigator to be related to the study intervention. Statistical analysis included only Groups 1 and 2 as indicated by the protocol.
Time Frame: Up to Day 35 (up to 14 days after completing study treatment)
Population: All participants in Groups 1, 2, and 3 who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 31 | 16 | 3
Percentage of Participants | 0.0 | 0.0 | 33.3
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in drug-related SAE % = 0.0, 95% CI 2-sided [-19.7 to 11.2] — Miettinen & Nurminen method

6. Primary Outcome: Percentage of Participants Discontinuing From Study Therapy Due to ≥1 AEs
Description: The percentage of participants in Group 1, 2, and 3 discontinuing from study drug due to ≥1 AEs during the treatment period was determined. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Statistical analysis included only Groups 1 and 2 as indicated by the protocol.
Time Frame: Up to Day 21
Population: All participants in Groups 1, 2, and 3 who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 31 | 16 | 3
Percentage of Participants | 0.0 | 18.8 | 33.3
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in discontinuation % = -18.8, 95% CI 2-sided [-43.3 to -6.2] — Miettinen & Nurminen method

7. Primary Outcome: Percentage of Participants Discontinuing From Study Therapy Due to ≥1 Drug-Related AEs
Description: The percentage of participants in Groups 1, 2, and 3 discontinuing from study drug due to ≥1 drug-related AEs during the treatment period was determined. A drug-related AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, and considered by the investigator to be related to the study intervention. Statistical analysis included only Groups 1 and 2 as indicated by the protocol.
Time Frame: Up to Day 21
Population: All participants in Groups 1, 2, and 3 who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 31 | 16 | 3
Percentage of Participants | 0.0 | 12.5 | 33.3
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in drug-related discon % = -12.5, 95% CI 2-sided [-36.3 to -0.3] — Miettinen & Nurminen method

8. Primary Outcome: Analysis of Specific AEs With an Incidence of ≥4 Participants in a Treatment Group
Description: The percentage of participants experiencing AEs that occurred in ≥4 participants within either Group 1 or Group 2 was assessed. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Statistical analysis included only Groups 1 and 2 as indicated by the protocol; Group 3 had <4 participants and therefore no data are presented.
Time Frame: Up to Day 35 (up to 14 days after completing study treatment)
Population: All participants in Groups 1 and 2 who received ≥1 dose of study drug are included. Group 3 data is not shown for this measure because there are only 3 participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 31 | 16 | 0
Percentage of Participants
  Pyrexia | 12.9 | 12.5 |
  Blood creatinine increased | 0.0 | 25.0 |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in pyrexia % = 0.4, 95% CI 2-sided [-25.2 to 19.7] — Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference blood creatinine inc % = -25.0, 95% CI 2-sided [-49.8 to -10.1] — Miettinen & Nurminen method

9. Primary Outcome: Percentage of Participants With ≥1 Events of Clinical Interest (ECI)
Description: The percentage of participants in Groups 1, 2, and 3 having ECIs within 2 categories was determined. Category 1 ECIs included post-baseline laboratory values of an elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value that is ≥3x upper limit of normal (ULN) and an elevated total bilirubin value that is ≥2x ULN and (at the same time) an alkaline phosphatase value that is ≤2x ULN. Category 2 ECIs included a confirmed elevated AST or ALT value that is ≥5x ULN. Statistical analysis included only Groups 1 and 2 as indicated by the protocol.
Time Frame: Up to Day 35 (up to 14 days after completing study treatment)
Population: All participants in Groups 1, 2, and 3 who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 31 | 16 | 3
Percentage of Participants
  Category 1 ECI: number analyzed (Participants) | 31 | 16 | 0
  Category 1 ECI | 0.0 | 12.5 |
  Category 2 ECI: number analyzed (Participants) | 31 | 16 | 0
  Category 2 ECI | 0.0 | 12.5 |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in Category 1 ECI %; p = 0.047, Miettinen and Nurminen method; Difference in Category 1 ECI % = -12.5, 95% CI 2-sided [-36.3 to -0.3]
Statistical Analysis 2: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in Category 2 ECI %; p = 0.047, Miettinen and Nurminen method; Difference in Category 2 ECI % = -12.5, 95% CI [-36.3 to -0.3]

10. Secondary Outcome: Percentage of Participants With ≥1 Events of Treatment-Emergent Nephrotoxicity
Description: Treatment-emergent nephrotoxity was assessed in Groups 1 and 2 as indicated by the protocol (Group 3 was not included). Nephrotoxicity for participants with normal baseline serum creatinine levels (<1.2 mg/dL) was defined as "doubling of serum creatinine to >1.2 mg/dL or reduction in creatinine clearance (ClCR) of ≥50%". Nephrotoxicity for participants with pre-existing renal dysfunction (baseline serum creatinine level ≥1.2 mg/dL) was defined as "increase in serum creatinine by ≥1 mg/dL or reduction from baseline ClCR of ≥20% or need for renal replacement therapy (RRT)".
Time Frame: Up to Day 35 (up to 14 days after completing study treatment)
Population: All participants in Groups 1 and 2 who received ≥1 dose of study drug are included. Per protocol, Group 3 was not included in the nephrotoxicity analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 31 | 16 | 0
Percentage of Participants | 10.3 [2.8 to 27.2] | 56.3 [33.2 to 76.9] |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; p = 0.002, Fisher Exact; Difference in nephrotoxicity % = -45.9, 95% CI [-69.1 to -18.4] — Miettinen & Nurminen method

11. Secondary Outcome: Percentage of Participants With Favorable Clinical Response (FCR) at Day 28
Description: The percentage of participants with FCR at Day 28 was determined for Groups 1 and 2. FCR at Day 28 was defined as "sustained cure" or "cure". Sustained cure (for participants with "cure" response at the prior visit) was defined as "all pretherapy signs and symptoms of index infection resolved with no evidence of resurgence and no additional antibiotic therapy required, and (for cIAI participants) no unplanned surgical procedures or percutaneous drainage procedures have been performed". Cure (for participants with "improved" response at EOT visit) was defined as "all pretherapy signs and symptoms of index infection resolved or returned to preinfection status, and no additional IV antibiotic therapy required, and (for cIAI participants) no unplanned surgical procedures or percutaneous drainage procedures performed".
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 21 | 10 | 0
Percentage of Participants | 71.4 [49.8 to 86.4] | 40.0 [16.7 to 68.8] |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in Day 28 FCR %; Difference in Day 28 FCR % = 26.3, 90% CI 2-sided [1.3 to 51.5] — Miettinen and Nurminen method stratified by infection-site stratum

12. Secondary Outcome: Percentage of Participants With All-cause Mortality Up to Day 28
Description: The percentage of participants with all-cause mortality up to Day 28 was determined for Groups 1 and 2.
Time Frame: Up to Day 28
Population: Participants in Group 1 and Group 2 who received ≥1 dose of each trial drug within a given IV treatment regimen, and who had a baseline bacterial pathogen that met inclusion criteria, are included. As per protocol, efficacy data from open-label Group 3 was considered exploratory and not included in the comparative analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 21 | 10 | 0
Percentage of Participants | 9.5 [1.4 to 30.1] | 30.0 [10.3 to 60.8] |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in mortality %; Difference in mortality % = -17.3, 90% CI 2-sided [-46.4 to 6.7] — Miettinen and Nurminen method stratified by infection-site stratum

13. Secondary Outcome: Percentage of Participants With FCR on Therapy (OTX)
Description: The percentage of participants with a FCR at OTX was determined for Groups 1 and 2. FCR at OTX was defined as "improved". Improved was defined as "all or most pretherapy signs and symptoms of index infection have improved or resolved, and (for cIAI participants) no unplanned surgical procedures or percutaneous drainage procedures have been performed.
Time Frame: OTX (Day 3)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 21 | 10 | 0
Percentage of Participants | 81.0 [59.4 to 92.9] | 40.0 [16.7 to 68.8] |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Adjusted difference in OTX FCR %; Adjusted difference in OTX FCR % = 33.9, 90% CI 2-sided [7.4 to 61.1] — Miettinen and Nurminen method stratified by infection-site stratum

14. Secondary Outcome: Percentage of Participants With FCR at End of Therapy (EOT)
Description: The percentage of participants with FCR at EOT was determined for Groups 1 and 2. FCR at EOT was defined as "cure" or "improved". Cure was defined as "all pretherapy signs and symptoms of index infection resolved or returned to preinfection status, and no additional IV antibiotic therapy required, and (for cIAI participants) no unplanned surgical procedures or percutaneous drainage procedures performed". Improved was defined as "all or most pretherapy signs and symptoms of index infection have improved or resolved, and (for cIAI participants) no unplanned surgical procedures or percutaneous drainage procedures have been performed.
Time Frame: At EOT (up to Day 21)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 21 | 10 | 0
Percentage of Participants | 90.5 [69.9 to 98.6] | 60.0 [31.2 to 83.3] |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Adjusted difference in EOT FCR %; Adjusted difference in EOT FCR % = 25.4, 90% CI 2-sided [3.1 to 53.6] — Miettinen and Nurminen method stratified by infection-site stratum

15. Secondary Outcome: Percentage of Participants With FCR at EFU
Description: The percentage of participants with FCR at EFU was determined for Groups 1 and 2. FCR at EFU was defined as "sustained cure" or "cure". Sustained cure (for participants with "cure" response at the prior visit) was defined as "all pretherapy signs and symptoms of index infection resolved with no evidence of resurgence and no additional antibiotic therapy required, and (for cIAI participants) no unplanned surgical procedures or percutaneous drainage procedures have been performed". Cure (for participants with "improved" response at EOT visit) was defined as "all pretherapy signs and symptoms of index infection resolved or returned to preinfection status, and no additional IV antibiotic therapy required, and (for cIAI participants) no unplanned surgical procedures or percutaneous drainage procedures performed".
Time Frame: EFU (Between Day 10 and Day 30 [5 to 9 Days after EOT])
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 21 | 10 | 0
Percentage of Participants | 81.0 [59.4 to 92.9] | 50.0 [23.7 to 76.3] |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Adjusted difference in EFU FCR %; Difference in EFU FCR % = 24.7, 90% CI 2-sided [3.8 to 51.4] — Miettinen and Nurminen method stratified by infection-site stratum

16. Secondary Outcome: Percentage of cUTI Participants With Favorable Microbiological Response (FMR) at OTX
Description: The percentage of participants with FMR at OTX was determined for participants with cUTI in Groups 1 and 2. FMR was defined as "urine culture results at OTX showing eradication (i.e., ≥10^5 colony forming units [CFU]/mL at baseline was reduced to <10^4 CFU/mL at OTX) of the uropathogen".
Time Frame: OTX (Day 3)
Population: Participants in Group 1 and Group 2 with cUTI who received ≥1 dose of each trial drug within a given IV treatment regimen, and who had a baseline bacterial pathogen that met inclusion criteria, are included. As per protocol, efficacy data from open-label Group 3 was considered exploratory and not included in the comparative analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 11 | 5 | 0
Percentage of Participants | 100.0 [70.0 to 100.0] | 100.0 [51.1 to 100.0] |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in FMR % = 0.0, 90% CI 2-sided [-20.8 to 36.6] — Miettinen & Nurminen method

17. Secondary Outcome: Percentage of cUTI Participants With FMR at EOT
Description: The percentage of participants with FMR at EOT was determined for participants with cUTI in Groups 1 and 2. FMR was defined as "urine culture results at EOT showing eradication (i.e., ≥10^5 CFU/mL at baseline was reduced to <10^4 CFU/mL at EOT) or sustained eradication (i.e., ≥10^5 CFU/mL at baseline that was reduced to <10^4 CFU/mL previously remained <10^4 CFU/mL at EOT) of the uropathogen".
Time Frame: At EOT (up to Day 21)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 11 | 5 | 0
Percentage of Participants | 100.0 [70.0 to 100.0] | 100.0 [51.1 to 100.0] |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in FMR % = 0.0, 90% CI 2-sided [-20.8 to 36.6] — Miettinen & Nurminen method

18. Secondary Outcome: Percentage of cUTI Participants With FMR at EFU
Description: The percentage of participants with FMR at EFU was determined for participants with cUTI in Groups 1 and 2. FMR was defined as "urine culture results at EFU showing sustained eradication (i.e., ≥10^5 CFU/mL at baseline that was reduced to <10^4 CFU/mL previously remained <10^4 CFU/mL at EFU) of the uropathogen".
Time Frame: EFU (Between Day 10 and Day 30 [5 to 9 Days after EOT])
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
Number analyzed (Participants) | 11 | 5 | 0
Percentage of Participants | 72.7 [42.9 to 90.8] | 100.0 [51.1 to 100.0] |
Statistical Analysis 1: Comparison: Group 1: Imipenem+Cilastatin/Relebactam vs Group 2: Colistimethate Sodium + Imipenem+Cilastatin; Test type: Other — Difference in percentages; Difference in FMR % = -27.3, 90% CI 2-sided [-52.8 to 12.8] — Miettinen & Nurminen method

ADVERSE EVENTS:
Time Frame: Up to Day 35 (up to 14 days after EOT)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. All participants in Groups 1, 2, and 3 who received ≥1 dose of study drug are included. Any event(s) reported to the investigator outside the AE monitoring period are also included.
Arm/Group | Group 1: Imipenem+Cilastatin/Relebactam | Group 2: Colistimethate Sodium + Imipenem+Cilastatin | Group 3: Open-Label Imipenem+Cilastatin/Relebactam
All-Cause Mortality (participants affected / at risk) | 2/31 | 3/16 | 1/3
Serious Adverse Events (participants affected / at risk) | 4/31 | 5/16 | 3/3
Other Adverse Events (participants affected / at risk) | 15/31 | 13/16 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Imipenem+Cilastatin/Relebactam (N=31) | Group 2: Colistimethate Sodium + Imipenem+Cilastatin (N=16) | Group 3: Open-Label Imipenem+Cilastatin/Relebactam (N=3)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic haematoma (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Imipenem+Cilastatin/Relebactam (N=31) | Group 2: Colistimethate Sodium + Imipenem+Cilastatin (N=16) | Group 3: Open-Label Imipenem+Cilastatin/Relebactam (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Infusion site phlebitis (General disorders) | 1 (1) | 2 (2) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (5) | 2 (2) | 0 (0)
Hepatic artery stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Periportal oedema (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Anorectal infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial abdominal infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Biliary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Biliary tract infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Peritoneal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory moniliasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Serratia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 4 (4) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Tracheal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT02452047/Prot_SAP_000.pdf